CLINICAL TRIAL: NCT05454475
Title: Effect of Different Water Injection Temperatures on the Safety and Comfort of Patients Undergoing Ultrasound Endoscopy of Small Probes Under Intravenous Anesthesia
Status: Completed | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Tian, MD, associate professor, The Third Xiangya Hospital of Central South University
Other Study IDs: fu3tianli
Record Dates: First submitted 2022-06-12; First posted 2022-07-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2022-07

CONDITIONS: Small Probe Ultrasound Endoscopy; The Water Temperature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low temperature group: The temperature is 6℃-10℃.
  Interventions: Other: Change the water injection temperature
- room temperature group: The temperature is 20℃-24℃.
  Interventions: Other: Change the water injection temperature
- Core temperature group: The temperature is 35℃-39℃.
  Interventions: Other: Change the water injection temperature

INTERVENTIONS:
Other: Change the water injection temperature — Water injection is a routine procedure for endoscopy of small probe ultrasound, and our intervention is to change the water temperature and observe the effects of different water temperatures on patient safety and comfort.

SUMMARY:
Miniprobe endoscopic ultrasonography (mEUS) is a key diagnostic modality for gastrointestinal (GI) mucosal or submucosal lesions, requiring water infusion to eliminate intraluminal air and improve image clarity. However, the optimal water temperature for sedated mEUS remains uncertain-previous studies suggest water temperature may affect GI peristalsis, haemodynamics, image quality, and patient safety/comfort, but no research has focused on this topic in sedated mEUS.

This is a prospective, multicentre, double-blind, randomized controlled study. Eligible patients (≥18 years with GI mucosal/submucosal lesions requiring sedated mEUS) are randomly assigned to three groups based on water temperature: cold water (6-10 °C), warm water (20-24 °C), and hot water (35-39 °C). The primary objectives are to evaluate the effects of different water temperatures on mEUS image quality (standardized scoring) and diagnostic accuracy. Secondary outcomes include GI peristaltic grade, haemodynamic indices (measured at 6 time points), adverse events, and patient somatic/psychological feeling, comfort, and satisfaction scores.

The study aims to identify the optimal water temperature that reduces GI peristalsis, improves mEUS diagnostic performance, and ensures patient safety and comfort during sedated mEUS, providing evidence for standardized clinical practice.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years old;
* Gastrointestinal (GI) mucosal or submucosal lesions detected by general endoscopy;
* Require small-probe ultrasonic endoscopy (mEUS) under sedation for definitive diagnosis;
* Clearly understand the study and voluntarily participate, with informed consent provided.

Exclusion Criteria

* Failure to meet the requirements for mEUS examination and anaesthesia, or need to use multiple sedative and analgesic drugs;
* Pregnancy or breastfeeding;
* Chronic use of opioids and benzodiazepines;
* Structural changes in the GI tract caused by abdominal surgery;
* Presence of mental illness;
* Presence of lesions in the oesophagus.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In the Third Xiangya Hospital of Central South University, the First Affiliated Hospital of South China University, the South China Hospital Affiliated to the University of South China, the Hunan Provincial People's Hospital, and the First People's Hospital of Changde City, patients with small probe ultrasound endoscopy under intravenous anesthesia due to gastrointestinal bulge lesions.
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
mEUS image quality | From examination initiation through 24 hours post-examination
  Assessed by two independent experts (excluding the operating endoscopist) using Soon's scoring method on a 1-5 scale: 1 = air artifact obscures target lesion; 2 = air artifact severely impairs lesion size/characteristic assessment; 3 = air artifact mildly impairs lesion size/characteristic assessment; 4 = air artifact present but does not compromise lesion assessment; 5 = no air artifact with unimpaired lesion assessment. Scores 1-2 = poor, 3-4 = good, 5 = excellent.
mEUS diagnostic accuracy | Up to 6 months after mEUS examination
  Gold standard confirmation: surgical, ESD or puncture histopathological results for patients with tissue specimens; ≥6-month clinical follow-up (based on manifestations, test results, lesion size and echogenic changes) for determining benign/malignant nature in other patients.

SECONDARY OUTCOMES:
Gastrointestinal (GI) peristaltic grade | During mEUS examination
  Assessed by two independent experts (excluding the operating endoscopist) via recorded video, using Hiki's upper GI peristaltic score and Likman Mui's lower GI peristaltic score (1=no peristalsis; 5=markedly vigorous peristalsis).
Haemodynamic indices | At T0, T1, T2, T3, T4, and T5 time points
  Includes mean arterial pressure (MAP), heart rate (HR), and oxygen saturation (SpO2); measured at 6 time points: anaesthesia assessment (T0), endoscopy (T1), before water infusion (T2), at water infusion (T3), after total water aspiration (T4), and at wakefulness (T5).
Adverse events | Periprocedural (from anesthesia assessment to post-anesthesia wakefulness)
  Includes coughing, choking, aspiration, hypotension (MAP during/after water infusion <20% of pre-infusion level), bradycardia (HR <50 beats/min), tachycardia (HR >100 beats/min), hypoxaemia (SpO2 <90%), bleeding, perforation, and infection.
Somatic and psychological feeling scores | Post-anesthesia recovery (Day 1)
  Assessed via questionnaire post-anesthesia recovery: somatic discomfort (nausea/vomiting, bloating, coldness, anxiety); pain (VAS: 0=no pain to 10=severe pain); comfort and satisfaction (5-point Likert scale: 1=very uncomfortable/dissatisfied to 5=very comfortable/satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: L Tian, Study Chair — The Third Xiangya Hospital of Central South University
Locations (1):
- he Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.